CLINICAL TRIAL: NCT03172013
Title: Platelet Indices Could Predict Spontaneous Bacterial Peritonitis in Cirrhotic Ascitic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Sponsor
Other Study IDs: eldemerdash
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cirrhotic ascitic patients with SBP,: Cirrhotic ascitic patients with SBP,
  Interventions: Diagnostic Test: Platelet indices
- cirrhotic ascitic patients without SBP,: cirrhotic ascitic patients without SBP,
  Interventions: Diagnostic Test: Platelet indices
- Healthy volunteers: Healthy individuals
  Interventions: Diagnostic Test: Platelet indices

INTERVENTIONS:
Diagnostic Test: Platelet indices — MPV, PDW

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is an ascitic fluid infection in cirrhotic patients

DETAILED DESCRIPTION:
Platelet indices can be utilized as a non-invasive predictor of SBP.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients and ascites

Exclusion Criteria:

* patients with ascites due to causes other than cirrhosis- immunocompromised patients,
* patients with abnormal thrombocytes due to non-hepatic causes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cirrhotic ascites
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with SBP and abnormal platelet indices | 6 months
  Number of patients with SBP and abnormal platelet indices

CONTACTS AND LOCATIONS:
Overall Officials: Taher Eldemerdash, Professor, Principal Investigator — Consultant of Hepatology - Tanta University
Locations (1):
- Tanta university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided